CLINICAL TRIAL: NCT03214549
Title: Marginal Adaptation of E.Max Laminate Veneers Prepared With Modified Gull Wing Preparation and Conventional Preparation
Brief Title: Comparison in Marginal Adaptation Between Conventional and Gull Wing Preparation in Laminates Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Housham nabiel hassan musa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoUni
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Teeth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gull wing preparation veneers (Active Comparator): intervention: gull wing preparation in laminates veneers proximal margin of the preparation is placed toward the lingual .The area of the proximal margin between the contact area and the gingival papilla is placed even further to the lingual. This preparation design helps to hide the margin when the restorations are viewed from an angle.
  Interventions: Procedure: gull wing preparation of laminates veneers
- conventional preparation veneers (Active Comparator): intervention: conventional preparation in laminates veneers preparation of veneers without lingual extension of preparation in mesial and distal areas
  Interventions: Procedure: conventional preparation of laminates veneers

INTERVENTIONS:
Procedure: gull wing preparation of laminates veneers — preparation involving mesial and distal extension further lingualy.
  Other Names: dog leg preparation of laminates veneers
  Arms: gull wing preparation veneers
Procedure: conventional preparation of laminates veneers — preparation not involving mesial and distal extension further lingualy.
  Arms: conventional preparation veneers

SUMMARY:
The aim of this study is to evaluate tooth sensitivity and marginal adaptation of porcelain laminates veneers prepared with modified gull wing preparation and conventional preparation.

DETAILED DESCRIPTION:
Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radio-graphic examination and primary impression for diagnostic cast construction.

Visit 2: Teeth preparation, secondary impression,temporary restoration and teeth sensitivity evaluation using United States Public Health Service criteria.

Visit 3: Placement and permanent cementation of the final restoration

Visit 4: marginal adaptation measurement by electron microscope using impression replica.

ELIGIBILITY:
Inclusion Criteria:

* From 18-40 years old, be able to read and sign the informed consent document.
* Be physically and psychologically able to tolerate conventional restorative Procedures.
* Have no active periodontal or pulpal diseases, have teeth with good restorations.
* Patients with teeth problems indicated for laminate veneer (e.g:discoloration, fracture not involve more than 50% enamel loss, mild malposition.
* Be willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth.
* Patient with fractured teeth of more than 50% enamel loss.
* Patients with poor oral hygiene and motivation.
* Pregnant women.
* Patient with post and core endodontically treated teeth.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for restoration

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-07-13 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
measuring marginal adaptation of laminates veneers using stero-microscope | immediately before laminates delivery up to 4 week sfter tooth preparation
  marginal adaptation of laminates veneers will be assess as follows, before laminates cementation, an impression material will be placed in the fitting surface of the veneers and placed over the reduced tooth using finger pressure, after material set the impression replica is separated from the laminates and the replica is section and measures under stero-microscope for marginal adaptation, measurement will be performed in eight different points on the buccal and mesio-distal sections, measurement will be in micrometer.

SECONDARY OUTCOMES:
measuring tooth sensitivity after tooth preparation for laminates veneers | one week after tooth preparation
  measurment will be acording tomodified United States Public Health Service (USPHS) criteria used for the clinical evaluations of the restorations. post-operative sensitivity 0 No symptoms
  1. Slight sensitivity
  2. Moderate sensitivity
  3. Severe pain

IPD SHARING:
Plan to Share IPD: Undecided